CLINICAL TRIAL: NCT02261298
Title: ONO-4538 Multicenter, Open-label, Uncontrolled, Phase I Multiple Dose Study in Solid Tumor
Brief Title: ONO-4538 Phase I Study in Patients With Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONO-4538-14
Record Dates: First submitted 2014-09-30; First posted 2014-10-10 (Estimated); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Advanced Solid Tumors; Recurrent Solid Tumors
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ONO-4538 1mg/kg (Experimental): ONO-4538 water-soluble injection, 100 mg/vial, 1mg/kg, 3 times once every 2 weeks in each 6-week cycle
  Interventions: Drug: ONO-4538
- ONO-4538 3mg/kg (Experimental): ONO-4538 water-soluble injection, 100 mg/vial, 3mg/kg, 3 times once every 2 weeks in each 6-week cycle
  Interventions: Drug: ONO-4538
- ONO-4538 10mg/kg (Experimental): ONO-4538 water-soluble injection, 100 mg/vial, 10mg/kg, 3 times once every 2 weeks in each 6-week cycle
  Interventions: Drug: ONO-4538

INTERVENTIONS:
Drug: ONO-4538

SUMMARY:
The objective of this study is to investigate the safety, pharmacokinetics, pharmacology and efficacy of ONO-4538 administered to Korean patients with advanced or recurrent solid tumors who are refractory or intolerant to standard therapy or for whom no appropriate treatment is available.

ELIGIBILITY:
Inclusion Criteria:

* The treatment phase has been completed in the ONO-4538-13 study

Exclusion Criteria:

* The development of PD is identified by the principal or sub investigator according to the RECIST guideline (version 1.1) only in case in which the unplanned tumor assessment with diagnostic image is performed in the treatment phase of ONO-4538-13 study.
* It is determined that continuing the treatment is not appropriate because the worsening of clinical symptoms attributed to disease progression occurs.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Safety outcome: The number of subjects with overall adverse events | Approximately 6 months
Safety outcome: The number of deaths | Approximately 6 months
PK outcome: Cmax of ONO-4538 | Approximately 10 months
Efficacy outcome: Response rate | Approximately 6 months
Efficacy outcome: Progression free survival | Approximately 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mitsunobu Tanimoto, Study Director — Ono Pharmaceutical Co. Ltd
Locations (5):
- South Korea (5):
  - Seongnam-si Clinical Site 105, Seongnam-si, Gyeonggi-do
  - Seoul Clinical Site 101, Seoul
  - Seoul Clinical Site 102, Seoul
  - Seoul Clinical Site 103, Seoul
  - Seoul Clinical Site 104, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee KW, Lee DH, Kang JH, Park JO, Kim SH, Hong YS, Kim ST, Oh DY, Bang YJ. Phase I Pharmacokinetic Study of Nivolumab in Korean Patients with Advanced Solid Tumors. Oncologist. 2018 Feb;23(2):155-e17. doi: 10.1634/theoncologist.2017-0528. Epub 2017 Nov 20. PMID 29158363